CLINICAL TRIAL: NCT04394299
Title: Cognitive Impairment and Clinical Characteristics in Patients With Chronic Obstructive Pulmonary Disease: Retrospective Study
Brief Title: Cognitive Impairment in COPD Patients
Acronym: RESCOG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Dr. Patrizia Russo, Principal Investigator, IRCCS San Raffaele
Other Study IDs: IRCCSSanRaffaele
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: COPD
Keywords: COPD; Cognitive impairment; Pulmonary rehabilitation; Outcome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prior researches suggest the presence of impaired lung function may be linked to cognitive impairment (CI). A recent study shows that lung disease, and specifically Chronic obstructive pulmonary disease (COPD) are associated to a greater risk of CI in a population of 14,184 individuals followed for over 23 years. Moreover, the study shows that low forced expiratory volume in 1 second (FEV1) is associated to an increased risk of dementia and MCI, indipendently of smoking habit.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is considered "a progressive but potentially treatable and preventable disease". The clinical view of COPD is moved from a lung-centered model to a novel one that considers COPD as an "umbrella" term encompassing different pulmonary and extra-pulmonary manifestations.

Prior researches suggest the presence of impaired lung function may be linked to cognitive impairment (CI). Among these studies, one prospective found that a diagnosis of COPD is associated with an increased risk of mild cognitive impairment (MCI), mainly nonamnestic MCI (NA-MCI), in a dose-response relationship between COPD duration and risk of MCI. Moreover, CI associated with severe COPD stage increases mortality. Among these studies only one shows that CI decreases adherence to pharmacological and non-pharmacological therapies. However, while it is well known that an MMSE score of 23-24 points or less is predictive of poor inhaler technique no studies report the impact of CI on PR outcomes. It has been reported that patients with MMSE < 24 walk lesser, at the basal level, than patients with a MMSE score > 24 (146 ±134 versus 242 ± 152 m) in the six minutes walking tests (6MWT) but no data are reported after rehabilitation. On the other hand, some papers report an association between participation in exercise rehabilitation programs and enhanced performance on cognitive tests.

The aim of this study is to compare cognitive functioning in patients with COPD referred for pulmonary rehabilitation to the response of the programme itself. More specific objectives of the present study are to:

* Study whether and to what extent CI in patients with COPD impacts outcomes of pulmonary rehabilitation such as 6MW distance (6MWD), Barthel and Borg scales for assessing dyspnea, Maugeri Foundation Respiratory Failure Questionnaire and the disease-specific respiratory quality of life (QoL) [St. George's Respiratory Questionnaire (SGRQ) and the Medical Research Council (MRC)].
* Investigate clinical and demographic characteristics of patients with COPD with cognitive impairment.

The hypothesize is that COPD patients with CI have worse response to PR compared with patients with no CI.

These results are important on the light of a personalized approach according to the so called "P4 medicine", for predictive, preventive, personalized and participatory Recently, the so-called "Rehabilomics" research framework, initially introduced r in traumatic brain injury rehabilitation, was applied on COPD rehabilitation. The "Rehabilomics" represents an exclusive and distinctive model in the path of the personalized-medicine approaches to rehabilitation. Thus, in previousstudy the Rehabilomics-like approach was used to afford the complexity of COPD rehabilitation, incorporating social/demographic data (i.e. gender, education, presence of a caregiver) clinical, psychological/emotional traits, genetics (i.e. DNA variants) and biological factors (i.e. DNA damage, levels of interleukins, et cet.) in a real life setting.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted consecutively

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with moderate to very severe diagnosis of COPD, based on GOLD criteria [Global Initiative for Chronic Obstructive Lung Disease. Report 2020 https://goldcopd.org/wp-content/uploads/2019/11/GOLD-2020-REPORT-ver1.0wms.pdf], who were admitted to inpatient clinic for a period of 3-4 weeks of comprehensive interdisciplinary pulmonary rehabilitation (PR) program from January 2012 to December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 1476 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive impairment | 2 months
  Mini Mental State Evaluation score from zero to 30
Response to Pulmonary Rehabilitation | 3 months
  Evaluation using six minutes walking test

SECONDARY OUTCOMES:
Evaluation of responders according to six minutes walking test | 3 months
  Patients able to walk for more of 30 meter after rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Russo, PhD, Principal Investigator — IRCCSSanraffaele
Locations (1):
- IRCCSSanraffaele, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vanfleteren LEGW, Spruit MA, Wouters EFM, Franssen FME. Management of chronic obstructive pulmonary disease beyond the lungs. Lancet Respir Med. 2016 Nov;4(11):911-924. doi: 10.1016/S2213-2600(16)00097-7. Epub 2016 Jun 2. PMID 27264777
- [Background] Prinzi G, Santoro A, Lamonaca P, Cardaci V, Fini M, Russo P. Cognitive Impairment in Chronic Obstructive Pulmonary Disease (COPD): Possible Utility of Marine Bioactive Compounds. Mar Drugs. 2018 Sep 4;16(9):313. doi: 10.3390/md16090313. PMID 30181485
- [Background] Yohannes AM, Chen W, Moga AM, Leroi I, Connolly MJ. Cognitive Impairment in Chronic Obstructive Pulmonary Disease and Chronic Heart Failure: A Systematic Review and Meta-analysis of Observational Studies. J Am Med Dir Assoc. 2017 May 1;18(5):451.e1-451.e11. doi: 10.1016/j.jamda.2017.01.014. Epub 2017 Mar 11. PMID 28292570
- [Background] Singh B, Mielke MM, Parsaik AK, Cha RH, Roberts RO, Scanlon PD, Geda YE, Christianson TJ, Pankratz VS, Petersen RC. A prospective study of chronic obstructive pulmonary disease and the risk for mild cognitive impairment. JAMA Neurol. 2014 May;71(5):581-8. doi: 10.1001/jamaneurol.2014.94. PMID 24637951
- [Background] Cleutjens FA, Janssen DJ, Ponds RW, Dijkstra JB, Wouters EF. COgnitive-pulmonary disease. Biomed Res Int. 2014;2014:697825. doi: 10.1155/2014/697825. Epub 2014 Mar 16. PMID 24738069
- [Background] Cleutjens FAHM, Spruit MA, Ponds RWHM, Vanfleteren LEGW, Franssen FME, Gijsen C, Dijkstra JB, Wouters EFM, Janssen DJA. Cognitive impairment and clinical characteristics in patients with chronic obstructive pulmonary disease. Chron Respir Dis. 2018 May;15(2):91-102. doi: 10.1177/1479972317709651. Epub 2017 May 29. PMID 28553720
- [Background] Pierobon A, Sini Bottelli E, Ranzini L, Bruschi C, Maestri R, Bertolotti G, Sommaruga M, Torlaschi V, Callegari S, Giardini A. COPD patients' self-reported adherence, psychosocial factors and mild cognitive impairment in pulmonary rehabilitation. Int J Chron Obstruct Pulmon Dis. 2017 Jul 18;12:2059-2067. doi: 10.2147/COPD.S133586. eCollection 2017. PMID 28790808
- [Background] Pierobon A, Ranzini L, Torlaschi V, Sini Bottelli E, Giardini A, Bruschi C, Maestri R, Callegari S, Raccanelli R, Sommaruga M. Screening for neuropsychological impairment in COPD patients undergoing rehabilitation. PLoS One. 2018 Aug 1;13(8):e0199736. doi: 10.1371/journal.pone.0199736. eCollection 2018. PMID 30067787
- [Background] Baird C, Lovell J, Johnson M, Shiell K, Ibrahim JE. The impact of cognitive impairment on self-management in chronic obstructive pulmonary disease: A systematic review. Respir Med. 2017 Aug;129:130-139. doi: 10.1016/j.rmed.2017.06.006. Epub 2017 Jun 15. PMID 28732820
- [Background] Ozyemisci-Taskiran O, Bozkurt SO, Kokturk N, Karatas GK. Is there any association between cognitive status and functional capacity during exacerbation of chronic obstructive pulmonary disease? Chron Respir Dis. 2015 Aug;12(3):247-55. doi: 10.1177/1479972315589748. Epub 2015 Jun 11. PMID 26071384
- [Background] Emery CF, Schein RL, Hauck ER, MacIntyre NR. Psychological and cognitive outcomes of a randomized trial of exercise among patients with chronic obstructive pulmonary disease. Health Psychol. 1998 May;17(3):232-40. doi: 10.1037//0278-6133.17.3.232. PMID 9619472
- [Background] Hood L, Flores M. A personal view on systems medicine and the emergence of proactive P4 medicine: predictive, preventive, personalized and participatory. N Biotechnol. 2012 Sep 15;29(6):613-24. doi: 10.1016/j.nbt.2012.03.004. Epub 2012 Mar 18. PMID 22450380
- [Background] Wagner AK. TBI Rehabilomics Research: an Exemplar of a Biomarker-Based Approach to Precision Care for Populations with Disability. Curr Neurol Neurosci Rep. 2017 Sep 19;17(11):84. doi: 10.1007/s11910-017-0791-5. PMID 28929311